CLINICAL TRIAL: NCT01400165
Title: Examination of the Pharmacokinetic Properties of Three Generic Medications and Their Respective Brand Preparations in Healthy Male Volunteers
Brief Title: Comparison of the Pharmacokinetics of Three Generic Medications and Their Respective Brand Preparations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Dr Pierre BLIER, MD, PhD, University of Ottawa, Institute of Mental Health Research - Mood Disorders Research Unit
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB-2010023
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: Therapeutic Equivalency; Human Experimentation; Bioequivalence; Brand name; Generic; Healthy volunteers
MeSH Terms: interventions — Trazodone; Quetiapine Fumarate; Pindolol; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desyrel/Teva-Trazodone (Active Comparator): Both drugs will be given at the dose of 150 mg. A washout period (corresponding to 10 half-life of the active compound) will be respected after receiving each medication.
  Interventions: Drug: Trazodone; Procedure: Blood Collection
- Visken/Teva-Pindolol (Active Comparator): Both drugs will be given at the dose of 10 mg. A washout period (corresponding to 10 half-life of the active compound) will be respected after receiving each medication
  Interventions: Drug: Pindolol; Procedure: Blood Collection
- Seroquel/Teva-Quetiapine (Active Comparator): Both drugs will be given at the dose of 100 mg. A washout period (corresponding to 10 half-life of the active compound) will be respected after receiving each medication
  Interventions: Drug: Quetiapine; Procedure: Blood Collection

INTERVENTIONS:
Drug: Trazodone — each subject will be taken 1 tablet of Trazodone 150mg of each group (brand/generic)
  Other Names: Desyrel; Teva-Trazodone
  Arms: Desyrel/Teva-Trazodone
Drug: Quetiapine — each subject will be taken 1 tablet of Quetiapine 100mg of each group (brand/generic)
  Other Names: Seroquel; Teva-Quetiapine
  Arms: Seroquel/Teva-Quetiapine
Drug: Pindolol — each subject will be taken 1 tablet of Pindolol 10mg of each group (brand/generic)
  Other Names: Visken; Teva-Pindolol
  Arms: Visken/Teva-Pindolol
Procedure: Blood Collection — Blood Samples will be collected at a predefined time-frame to study the plasma level of each medication.

SUMMARY:
Generic describes a pharmaceutical product that does not have a brand name or trademark. Generic medications should be the equivalent of brand medications. Only their price should be different. The active ingredient of the generic medication has to be within a window of 80 to 125% of the original in the blood. There are reports that this standard is not always followed after the medication has been on the market. Indeed, it was observed that some patients previously stable on original medications relapsed when switched to a generic. Several factors could account for this problem. Such problems have been reported for Pindolol, Quetiapine, and Trazodone. Some properties of specific brands of the generics and the original brands will be examined for these three medications. The three original medications used in this study are the Visken, the Seroquel, and the Desyrel. The three generics are the Teva-pindolol, the Teva-Quetiapine, and the Teva-Trazodone. They are all available on the Canadian market by prescription.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (absence of diseases: psychiatric, physical, neurological, metabolic,...)

Exclusion Criteria:

* Psychiatric disorder
* Hepatic disease
* Renal disease
* Gastrointestinal disease
* Hematological disease
* Smokers
* Physical and/or neurological disease
* Positive urine drug screen
* Abnormal blood pressure
* Abnormal Electrocardiogram
* Abnormal urine/blood analysis (sodium, potassium, chloride, creatinine, urea, ALT, AST, total protein, glucose, and TSH)
* Taking medication
* Have donated 50 mL to 499 mL whole blood within 30 days and more than 499 mL whole blood within 56 days preceding entry into this study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of Medication | 0 to 48 hours after drug ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Blier, MD, PhD, Principal Investigator — University of Ottawa, Institute of Mental Health Research - Mood Disorders Research Unit; Franck Chenu, PharmD, Phd, Principal Investigator — University of Ottawa, Institute of Mental Health Research - Mood Disorders Research Unit
Locations (1):
- University of Ottawa, Institute of Mental Health Research, Ottawa, Ontario, Canada